CLINICAL TRIAL: NCT03954743
Title: A Phase III, Observer-blind, Randomized, Multi-country Study to Assess the Reactogenicity and Safety of the Porcine Circovirus (PCV) Free Liquid Formulation of GSK's Oral Live Attenuated Human Rotavirus (HRV) Vaccine as Compared to the Lyophilized Formulation of the GSK's HRV Vaccine, When Administered as a 2-dose Vaccination in Infants Starting at Age 6-12 Weeks
Brief Title: Safety Study of 2 Formulations of GSK's Human Rotavirus (HRV) Vaccine (444563), in Healthy Infants Starting at Age 6-12 Weeks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 208236; 2018-001986-18 (EudraCT Number)
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Infections, Rotavirus
Keywords: HRV; Lyophilized formulation; Liquid formulation; Human rotavirus vaccine; Rotarix; Healthy infants; PCV-free; Porcine circovirus-free
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data were collected in an observer-blind manner. By observer-blind, it is meant that during the study period, the vaccine(s) recipient and those responsible for the evaluation of any study endpoint (e.g. safety and reactogenicity) were all unaware of which vaccine was administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HRV PCV-free Liq Group (Experimental): Subjects aged 6 to 12 weeks at the time of first vaccination, who received two doses of oral live-attenuated human rotavirus (HRV) porcine circovirus (PCV)-free vaccine in liquid formulation, one at Day 1 and one at Month 1 or Month 2, according to the immunization schedule for rotavirus (RV) vaccine administration in participating countries. PCV-free implies no detection of PCV-1 and PCV-2 according to the limit of detection of the tests used.
  Interventions: Biological: PCV-free liquid formulation of GSK's oral live attenuated HRV vaccine
- HRV Lyo group (Active Comparator): Subjects aged 6 to 12 weeks at the time of first vaccination, who received two doses of oral live-attenuated human rotavirus (HRV) vaccine in lyophilized formulation, one at Day 1 and one at Month 1 or Month 2, according to the immunization schedule for rotavirus (RV) vaccine administration in participating countries.
  Interventions: Biological: Lyophilized formulation of GSK's oral live attenuated HRV vaccine

INTERVENTIONS:
Biological: PCV-free liquid formulation of GSK's oral live attenuated HRV vaccine — 2 doses administered orally at Day 1 and at Month 1 or Month 2, according to the immunization schedule for RV vaccine administration in participating countries.
  Arms: HRV PCV-free Liq Group
Biological: Lyophilized formulation of GSK's oral live attenuated HRV vaccine — 2 doses administered orally at Day 1 and at Month 1 or Month 2, according to the immunization schedule for RV vaccine administration in participating countries.
  Arms: HRV Lyo group

SUMMARY:
The purpose of this study is to complete the total safety database size for GlaxoSmithKline Biologicals' (GSK's) human rotavirus (HRV) vaccine across the Porcine circovirus (PCV)-free development plan.

This study used a purposely selected lot for PCV-free liquid HRV vaccine that is in the upper range of the usual release potencies. The PCV-free liquid HRV vaccine lots used were stored frozen in order to keep the titer stable until administration during the study.

As the liquid formulation of GSK's HRV vaccine is not licensed in the US, the lyophilized formulation of the vaccine was used as a control in all phase III studies as part of the PCV-free development plan.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy all the following criteria at study entry:

* Subjects' parent(s)/LAR(s) who, in the opinion of the investigator, can and will comply, with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* Written or witnessed/thumb printed informed consent obtained from the parent(s)/LAR(s) of the subject prior to performance of any study specific procedure.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* A male or female between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination.

Exclusion Criteria:

Medical conditions

* Uncorrected congenital malformation (such as Meckel's diverticulum) of the gastrointestinal tract that would predispose for Intussusception (IS).
* Very prematurely born infants (born ≤28 weeks of gestation).
* History of IS.
* Family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Hypersensitivity to latex.
* Major congenital defects or serious chronic illness, as assessed by the investigator.
* Previous confirmed occurrence of Rotavirus Gastroenteritis (RV GE).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of Severe combined immunodeficiency (SCID). Prior/Concomitant therapy
* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study vaccines during the period starting 30 days before the first dose of study vaccines (Day -29 to Day 1), or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of study vaccine administration, with the exception of the inactivated influenza vaccine, which is allowed at any time during the study, and other licensed routine childhood vaccinations.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Administration of immunoglobulins and/or any blood products from birth or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone ≥0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Previous vaccination against RV. Prior/Concurrent clinical study experience
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or medical device).

Other exclusions

• Child in care.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1351 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- United States (17):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Frederick, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, East Orange, New Jersey
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Fairfield, Ohio
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Draper, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Charlottesville, Virginia
- Canada (9):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec
- Hong Kong (2):
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- Taiwan (3):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Eskişehir
  - GSK Investigational Site, Izmir
  - GSK Investigational Site, Kayseri

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 5 countries/regions (Canada, Hong Kong, Taiwan, Turkey and United States).
Pre-assignment Details: All 1351 participants enrolled in the study, received a study vaccination and were included in the Exposed Set.
Period: Overall Study
Arm/Group | HRV PCV-free Liq Group | HRV Lyo Group
Started | 677 | 674
Completed | 653 | 657
Not Completed | 24 | 17
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 6 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — CONSENT WITHDRAWAL NOT DUE TO ADV. EVENT | 13 | 12
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HRV PCV-free Liq Group | HRV Lyo Group | Total
Number analyzed (Participants) | 677 | 674 | 1351
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 9.0 (1.5) | 9.0 (1.5) | 9.0 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 336 | 357 | 693
  Male | 341 | 317 | 658
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 2 | 1 | 3
  Asian | 302 | 301 | 603
  Black Or African American | 14 | 10 | 24
  Native Hawaiian Or Other Pacific Islander | 0 | 2 | 2
  Other, Not specified | 20 | 14 | 34
  White | 339 | 346 | 685

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited General Adverse Events (AEs) After the First Vaccination
Description: Assessed solicited general AEs were fever (defined as temperature ≥ 38.0°C/100.4°F, the preferred location for measuring temperature in this study being the oral cavity, the axilla and the rectum), irritability/fussiness, diarrhea (defined as passage of three or more looser than normal stools within a day), vomiting (defined as one or more episodes of forceful emptying of partially digested stomach contents ≥1 hour after feeding within a day), loss of appetite and cough/runny nose. Any = occurrence of AE regardless of intensity grade or relation to study vaccination.
Time Frame: During the 8-day follow-up period after the first vaccination (vaccines administered at Day 1)
Population: Analysis was performed on the Exposed set (ES), which included all subjects with at least one study vaccine administration documented and with the diary card completed after the first vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | HRV PCV-free Liq Group | HRV Lyo Group
Number analyzed (Participants) | 677 | 674
Participants
  Cough / Runny Nose, Any | 139 | 166
  Diarrhea, Any | 41 | 47
  Fever, ≥ 38.0°C | 27 | 21
  Irritability / Fussiness, Any | 431 | 428
  Loss of appetite, Any | 201 | 186
  Vomiting, Any | 113 | 122

2. Primary Outcome: Number of Subjects With Any Solicited General Adverse Events (AEs) After the Second Vaccination
Description: as for outcome 1
Time Frame: During the 8-day follow-up period after the second vaccination (vaccines administered at Month 1 or Month 2)
Population: Analysis was performed on the Exposed set (ES), which included all subjects with at least one study vaccine administration documented and with the diary card completed after the second vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | HRV PCV-free Liq Group | HRV Lyo Group
Number analyzed (Participants) | 663 | 657
Participants
  Cough / Runny Nose, Any | 147 | 145
  Diarrhea, Any | 28 | 36
  Fever, ≥ 38.0°C | 46 | 40
  Irritability / Fussiness, Any | 368 | 362
  Loss of appetite, Any | 170 | 168
  Vomiting, Any | 82 | 88

3. Primary Outcome: Number of Subjects With Any Unsolicited AEs
Description: An unsolicited AE is defined as any untoward medical occurrence in a clinical study subject, temporally associated with the use of a study treatment, whether or not considered related to the study treatment, and reported in addition to those solicited during the clinical study and any 'solicited' AE with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of AE regardless of intensity grade or relation to study vaccination.
Time Frame: During the 31-day follow-up period across doses (vaccines administered at Day 1 and at Month 1 or Month 2)
Population: Analysis was performed on the Exposed set (ES), which included all subjects with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | HRV PCV-free Liq Group | HRV Lyo Group
Number analyzed (Participants) | 677 | 674
Participants | 201 | 206

4. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization and/or results in disability/incapacity. Any = occurrence of SAE regardless of intensity grade or relation to study vaccination.
Time Frame: Throughout the study period (from Day 1 up to Month 7 or Month 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HRV PCV-free Liq Group | HRV Lyo Group
Number analyzed (Participants) | 677 | 674
Participants | 39 | 38

ADVERSE EVENTS:
Time Frame: Solicited AEs: During the 8-day (Day 1 to Day 8) follow-up period after each HRV vaccination. Unsolicited AEs: During the 31-day (Day 1 to Day 31) follow-up period after any HRV vaccination. SAEs: Throughout the study period (from Day 1 up to Month 7 or Month 8).
Arm/Group | HRV PCV-free Liq Group | HRV Lyo Group
All-Cause Mortality (participants affected / at risk) | 0/677 | 0/674
Serious Adverse Events (participants affected / at risk) | 39/677 | 38/674
Other Adverse Events (participants affected / at risk) | 591/677 | 571/674
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HRV PCV-free Liq Group (N=677) | HRV Lyo Group (N=674)
Osteogenesis imperfecta (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Scaphocephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Adenovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Citrobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterovirus infection (Infections and infestations) | 2 (2) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Exanthema subitum (Infections and infestations) | 3 (3) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (2) | 4 (5)
Gastroenteritis enteroviral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Human bocavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 2 (2)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 2 (2)
Picornavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 5 (5) | 2 (2)
Rhinovirus infection (Infections and infestations) | 1 (1) | 2 (2)
Roseola (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 6 (6)
Urinary tract infection (Infections and infestations) | 6 (6) | 4 (4)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ear canal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (6) | 1 (2)
Kawasaki's disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HRV PCV-free Liq Group (N=677) | HRV Lyo Group (N=674)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 2 (2) | 1 (1)
Buried penis syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abnormal faeces (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (10) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 61 (76) | 81 (100)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 7 (7)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 3 (3)
Haematochezia (Gastrointestinal disorders) | 2 (3) | 4 (4)
Infantile colic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infantile spitting up (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 7 (9) | 7 (8)
Vomiting (Gastrointestinal disorders) | 153 (198) | 170 (219)
Discomfort (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 2 (2)
Irritability postvaccinal (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 92 (103) | 70 (79)
Swelling (General disorders) | 1 (1) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 5 (6) | 4 (5)
Milk allergy (Immune system disorders) | 0 (0) | 3 (3)
Bronchiolitis (Infections and infestations) | 8 (8) | 9 (9)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Candida nappy rash (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3) | 7 (7)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 2 (2) | 3 (3)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 30 (31) | 22 (24)
Omphalitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 3 (4) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 8 (9) | 3 (3)
Otitis media acute (Infections and infestations) | 1 (1) | 3 (3)
Paronychia (Infections and infestations) | 0 (0) | 3 (3)
Pharyngitis (Infections and infestations) | 6 (7) | 2 (2)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pustule (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 47 (52) | 46 (53)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea barbae (Infections and infestations) | 1 (1) | 0 (0)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 26 (31) | 34 (35)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral rash (Infections and infestations) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 7 (7) | 9 (9)
Body temperature increased (Investigations) | 2 (2) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 290 (371) | 261 (361)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 2 (3)
Somnolence (Nervous system disorders) | 2 (3) | 5 (6)
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 512 (812) | 487 (796)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 241 (295) | 239 (323)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (12)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 16 (17) | 8 (8)
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 9 (9)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT03954743/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03954743/SAP_001.pdf